CLINICAL TRIAL: NCT03782961
Title: Evaluation of Perceived Effectiveness to Evaluate Viscosity of a Vaginal Moisturizer in Menopaused Women
Brief Title: Evaluation of Viscosity of a Vaginal Moisturizer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Farmoquimica S.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FE4 - HIDRAFEMME - PA - 010
Record Dates: First submitted 2018-12-18; First posted 2018-12-20 (Actual); Last update posted 2018-12-21 (Actual); Status verified 2018-12

CONDITIONS: Vaginal Dryness; Menopausal Women

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stand up (Experimental): After application of the product (sodium lactate and combination of polymers) will remain standing for 30 minutes
  Interventions: Device: sodium lactate and combination of polymers
- Lying down (Experimental): After application of the product (sodium lactate and combination of polymers) remained lying down with the legs stretched for 30 minutes;
  Interventions: Device: sodium lactate and combination of polymers

INTERVENTIONS:
Device: sodium lactate and combination of polymers — sodium lactate and combination of polymers (polycarbophil, carbomer and PVM / MA copolymer)

SUMMARY:
To evaluate the perception of viscosity of a vaginal moisturizer in postmenopausal women

DETAILED DESCRIPTION:
A unicentric, blind, non-comparative clinical study to prove the perceived efficacy of the research product.

It will be necessary 33 female research participants, aged between 45 and 70 years menopause with complaint of vaginal dryness.

The participant will remain in the study for one day, making use of the research product in the Research Center.

Participants will be divided into 2 groups so that each group observes the viscosity (flow) of the test product in a different anatomical position (lying down and standing) immediately after application of the product, after 15 and 30 minutes.

Participants will respond to a subjective assessment using a standardized questionnaire to capture possible feelings of discomfort during the study.

A gynecologist will be available to monitor the participants throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Menopausal participants for at least 6 months;
* Participants with complaints of vaginal dryness;
* Skin integrity in the region of product analysis;
* Agreement to comply the procedures of the trial and attend the clinic on the days and times determined for applications and / or evaluations;
* Understanding, agreement and signing of the Informed Consent Term.

Exclusion Criteria:

* Use of anti-inflammatory / immunosuppressive / antihistamine drugs up to 3 weeks prior to selection;
* Pathologies and / or active skin lesions (local and / or disseminated) in the evaluation area;
* Immunosuppression by drugs or active diseases;
* Decompensated endocrinopathies;
* Relevant clinical history or current evidence of alcohol or other drug abuse;
* known history or suspected intolerance to products of the same category;
* Intense sun exposure up to 15 days before evaluation;
* Gynecological treatment up to 4 weeks before evaluation;
* Other conditions considered by the researcher to be reasonable for disqualification of study participation.

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2019-01-14 (Estimated); Primary Completion 2019-01-25 (Estimated); Study Completion 2019-01-25 (Estimated)

PRIMARY OUTCOMES:
To evaluate subjectively the perceived viscosity change | Immediately after application, 15 and 30 minutes after application
  Perceived viscosity change of the research product from the point of view of the target public under normal conditions of use through a questionnaire